CLINICAL TRIAL: NCT00422266
Title: Effect of Omega -3 Fatty Acids Supplements and Plant Sterol Enriched Drink/Food on the Composite Risk Profile of Dyslipidemic Adults
Brief Title: Effect of Omega -3 Fatty Acids Supplements and Plant Sterol Enriched Food in Dyslipidemic Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Chronic Disease Control, India (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCDC-6980
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Fatty Acids, Omega-3; Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Omega 3 fatty acids and plant sterol enriched drink
Dietary Supplement: Omega 3 fatty acids and plant sterols — Capsules and Yoghurt based minidrink

SUMMARY:
The incidence of chronic degenerative diseases, especially cardiovascular disease (CVD), is high world over and especially in India. High blood cholesterol and triglyceride levels are known to be important risk factors for CVD. There is a strong body of evidence for the beneficial effects of plant sterols on blood total and LDL-cholesterol and omega-3 fatty acids from fish on blood triglycerides. However, the combined benefits of consuming both plant sterols and omega-3 fatty acids from fish oil on blood cholesterol and triglycerides has not been investigated previously, except in one study where the methodology used was not the most appropriate for testing such a combination. In addition, most studies on plant sterol efficacy realised so far were done in Western countries. The present study will investigate the efficacy of plant sterols and omega-3 fatty acids from fish oil on improving the cardiovascular risk profile of Indian adults with dyslipidemia.

It is expected that, after 4 weeks of intervention, men consuming both plant sterols and omega-3 fatty acids from fish oil will have a lower cardiovascular risk profile than men receiving only plant sterols or only fish oil or none of these dietary supplements.

DETAILED DESCRIPTION:
This study has a double-blind, placebo-controlled, randomized parallel (2 x 2 factorial) design with 3 experimental treatments and one control treatment. A two week run-in period will be observed during which all subjects will be given placebos for plant sterols. Thereafter the subjects will be randomly allocated to the 4 treatment groups for the intervention period of 4 weeks and will undergo baseline assessment of blood lipids, inflammatory and coagulation markers, anthropometry, lifestyle and dietary habits. The intervention period will be closed by repeating measurements of lipids, inflammatory and coagulation markers, anthropometry, lifestyle and diet. Participants are mildly hypercholesterolemic adult males (TC between 5.0-8.0 mmol/L), aged between 35-55 years who are employees of NTPC, Badarpur, New Delhi will be enrolled in the study.

The subjects will be randomly allocated to the four treatment groups (1 control and 3 experimental, 50 subjects per group) with the help of computer generated random number tables. In case of a surplus of volunteers, a lottery method of selection will be applied.

The active and control products will be almost identical with respect to taste and appearance and will only differ in coding. During the study, the treatment code of the products will be blinded and only known by a person not directly involved in the study. The subjects will only be identified by a unique identification code given to them at the time of filling their interview-schedules. All the information obtained from the subjects will be coded using this unique identification code. During the intervention period the key linking subject's names and codes will only be accessible to authorized staff.

For each subject the Investigator and Sponsor will each receive a blinded code envelope with details of treatment. In case of an emergency (e.g. Serious Adverse Event possibly related to treatments, or unexpected Adverse Events), the envelope can be opened to identify the treatment given to a subject. The Investigator and Sponsor will immediately inform each other about such de-blinding.

Randomization data are kept strictly confidential until the time of unblinding. Only after the blind review meeting of PI, Investigator and Sponsor, the randomization codes will be broken and made available for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 35-55 years.
* Total cholesterol (TC) between 5.0 - 8.0 mmol/L.
* Body Mass Index (BMI) is between 18-30 kg/m2.
* Willing to consume the intervention product.
* Willing to participate in the study and perform all measurements including. blood drawing, anthropometry, dietary assessment and questionnaires.
* Informed consent signed by subject.

Exclusion Criteria:

* Smokers (more than 10 cigarettes per day).
* Heavy drinker (more than 6 large pegs or 360 ml of 40% alcohol per week).
* Triglycerides > 4.0 mmol/L.
* Individuals with chronic degenerative disease(s) such as diagnosed heart disease, cancer, stroke, diabetes, chronic renal failure, gastrointestinal disease, metabolic diseases (eg. thyroid, pancreas) and people with a compromised GI function like after extensive bowel resections.
* Fasting blood glucose > 120mg/dl and glycosylated hemoglobin > 7.5%.
* Individuals on medication (e.g.: insulin, oral hypoglycemic drugs, beta blockers, steroids or lipid-lowering drugs) or dietary supplements known to alter lipid and/or glucose metabolism during the study, including plant sterol-enriched foods and fish oil supplements, or having used these substances in 3 months preceding the intervention period.
* Reported participation in another biomedical trial 3 months before the start of the study or during the study.
* Reported weight loss / gain (10% or more) during the last 6 months.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2006-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Changes in TC, LDL-C, HDL-C, Triglycerides, and Fasting blood glucose.

SECONDARY OUTCOMES:
Changes in LDL particle size, apo B, CRP and fibrinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Srinath Reddy, MD, DM, MSc,, Principal Investigator — Centre for Chronic Disease Control, India; Prabhakaran Dorairaj, MD, DM, MSc, Principal Investigator — Centre for Chronic Disease Control
Locations (1):
- National Thermal Power Corporation, Delhi, Badarpur, India